CLINICAL TRIAL: NCT01165437
Title: Validation of a Novel Oscillometric-Based Algorithm for Determination of the Ankle-Brachial Index
Status: Completed | Type: Observational
Sponsor: Summit Doppler Systems, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: David C. Jones, Summit Doppler Systems, Inc.
Other Study IDs: CCF IRB 10-513
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral; Arterial; Vascular
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected Arterial Disease: Patients with known or suspected arterial disease and patients screened using AHA/ACC criteria for P.A.D.
  Interventions: Device: Blood Pressure Measurement

INTERVENTIONS:
Device: Blood Pressure Measurement — Systolic blood pressures will be obtained from each limb using Doppler, oscillometric, and photoplethysmographic (PPG) modalities.

SUMMARY:
Peripheral arterial disease (PAD) is a highly prevalent medical condition. Patients with PAD are usually diagnosed on the basis of the ankle-brachial index. The ankle-brachial index is the ratio of ankle pressure to arm pressure after measurement of blood pressures in the arms and legs using a Doppler device. The need for dedicated equipment and trained personnel, along with the time required to perform the test, have been identified as barriers to widespread implementation of ankle-brachial index screening. The use of automated oscillometric devices for blood pressure measurement has been applied to leg pressure measurement and determination of the ankle-brachial index with variable success. It will be beneficial to investigate a reliable oscillometric-based procedure that can accurately measure leg pressures for the ankle-brachial index across the entire spectrum of PAD severity.

In a previous pilot study completed in 2009 (IRB 08-823), the investigators gathered data from N=60 subjects which allowed for mathematical analysis of oscillometric waveforms derived from the lower extremities as compared to Doppler-based measurements of blood pressure. We used signal processing analysis and regression techniques to develop a two-step algorithm which will allow for accurate interpretation of oscillometric waveforms in normal/mild vs. moderate/severely diseased limb and accurate calculation of ankle pressure across the spectrum of peripheral artery disease severity.

This proposed project will validate this novel oscillometric ABI algorithm in a population of patients who have been identified as at risk for PAD and for whom screening ABI has been recommended by multiple professional organizations (AHA/ACC and American Diabetes Association). Arm, ankle, and toe pressure measurements will be made in the supine position using Doppler, oscillometric methods, and a photoplethysmographic sensor. The ankle-brachial index and toe-brachial index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* At least 70 years of age
* At least 50 years of age with a history of diabetes mellitus or tobacco smoking (>100 cigarettes in their lifetime)
* Ambulatory Outpatient

Exclusion Criteria:

* Unable to give informed consent
* Unable to lie supine for at least 15 minutes
* Known non-compressible vessels on prior laboratory studies (ABI>1.3 on either side)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the non-invasive vascular laboratory or another outpatient clinic in the Heart and Vascular Institute at Cleveland Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States